CLINICAL TRIAL: NCT04271046
Title: STAR Caregivers - Virtual Training and Follow-up
Acronym: STAR-C-VTF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1347434; 1R01AG061926-01 (NIH)
Record Dates: First submitted 2019-04-16; First posted 2020-02-17 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease; Dementia; Caregiver Burnout
MeSH Terms: conditions — Alzheimer Disease; Dementia; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: The trial will use a parallel, two-arm, randomized trial design. Participants will be randomly assigned to the experimental intervention or control. Participants in the control condition will receive mailed material from the Alzheimer's Association, web links and template secure messages. Everyone will complete assessments at baseline, 8-weeks post-enrollment, and 6 months post-enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group- STAR-C-VTF (Experimental): This study will use a parallel, two-arm randomized trial design. Participants will be 100 Person-with-Dementia-Caregiver dyads in which the person with dementia lives at home and recently filled a new prescription for antipsychotic medication. The experimental intervention will combine three elements:
  * self-directed learning in which the caregiver will receive training materials delivered electronically through a web-based learning portal;
  * one orientation phone visit with a coach;
  * ongoing support from the coach via telephone and secure messaging in the web-portal.
  Participants will complete self-report assessments at baseline, 8-weeks post-enrollment, and 6 months post-enrollment. Automated medication and primary care utilization data will be collected throughout the 6 month study period.
  Interventions: Behavioral: STAR-C-VTF
- Control (Active Comparator): One orientation phone visit with a coach. Participants in the control condition will receive mailed material from the Alzheimer's Association, web links and template secure messages.
  Participants will complete self-report assessments at baseline, 8-weeks post-enrollment, and 6 months post-enrollment. Automated medication and primary care utilization data will be collected throughout the 6 month study period.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: STAR-C-VTF — 1. One 60 minute baseline orientation phone visit with a coach to get verbal consent for participation in the study and to acquaint the caregiver with the STAR-VTF components of good dementia care; distribute printed educational material (and links to same material online);
  2. Six 30-minute follow-up phone calls with the caregiver following each of the 6 learning modules to review STAR-VTF concepts, and further brainstorm strategies to modify identified activators and consequences with the objective of reducing behavioral symptoms;
  3. secure message support, as needed, with the coach to help with personalizing the STAR-VTF curriculum for up to 6 months.
  Arms: Experimental Group- STAR-C-VTF
Behavioral: Control — One 60 minute baseline orientation phone visit with a coach to get verbal consent for participation in the study. Controls will receive usual care from their primary care provider and/or psychiatrist. We will give participants an information package from the Alzheimer's Association including a list of resources. To assist with retention, and to measure responses to secure messages, we will send a template secure message to control dyads once per month in which we remind participants to contact their primary care provider if they have any issues with behavioral and psychological symptoms of dementia. Dyads in the attention control may receive information and training from their primary care provider and the Alzheimer's Association. This "attention control" is proposed to assess the additional impact of STAR-VTF above treatment as usual. Investigators do not intend to track non-study training receipt in the control arm.
  Arms: Control

SUMMARY:
This study evaluates the effectiveness of a caregiver outreach, training, and support program for caregivers of people with dementia who are using antipsychotic medication to manage agitation/aggression. The Investigators will conduct a randomized trial of the caregiver program compared to a control group to measure differences in caregiver burden and discontinuation of antipsychotic medication use. The results will help in expanding access to and delivery of empirically supported behavioral health services for caregivers and people with dementia.

DETAILED DESCRIPTION:
Alzheimer's Disease and related dementias (ADRD) are debilitating conditions affecting more than 5 million Americans in 2014. With aging of the population it is projected that 8.4 million people will be diagnosed with ADRD over the next 15 years and health care costs attributable to ADRD are projected to be more than 1.2 trillion by 2050. Behavioral and Psychological Symptoms of Dementia (BPSD) (anxiety, agitation, depression) are common and often involve aggressive behavior towards family caregivers (CG) in response to unmet needs, discomfort, or frustration. BPSD are disturbing and frequently lead to caregivers seeking medication to control patient symptoms. Antipsychotic use in persons with dementia (PWD) more than doubles mortality risk; however, many caregivers are willing to accept those risks. The Choosing Wisely Guidelines from the American Psychiatric Association and American Geriatrics Society both recommend against prescribing antipsychotics as a first-line treatment for BPSD. STAR-Caregivers is an efficacious first-line behavioral treatment, endorsed by the Administration on Aging, that involves caregiver training to manage BPSD. However, the program has not been implemented widely - partly due to the cost of the programs, difficulty conducting outreach, and modality of training (in person with written materials). Adequate caregiver training and commensurate reduction in caregiver burden are the mediators (mechanisms) the Investigators will engage in this Stage III trial to reduce BPSD and discontinue antipsychotic medication use by PWD.

The STAR-Caregivers program is an education, training, and support intervention demonstrated efficacious in reducing BPSD. The original program involved 8 face-to-face, in-home training sessions and 4 follow-up phone calls. The condensed version involves 4 in-home sessions with 2 phone follow-ups.18 Neither of these is feasible from a payer perspective. The investigators propose to test a self-directed, remote version called STAR-virtual training and follow-up (STAR-VTF) that leverages secure email within the member portal at Kaiser Permanente Washington to improve access to training, fidelity to the STAR principles, and to lower the cost of the program.

The investigators propose a Stage III trial to ascertain the feasibility and acceptability of STAR-VTF in which (a) caregiver training materials are delivered electronically and learning is self-directed, (b) caregivers have one orientation phone visit with a social worker and (c) where caregivers receive ongoing support from a social worker via telephone and secure messaging in the web-based member portal. Investigators will compare outcomes in the STAR-VTF group to an attention control group (mailed material, links to websites, and generic secure messages).

The specific aims are:

Aim 1: Assess the feasibility and acceptability of conducting caregiver outreach, training, and support via social workers including: (1) willingness of caregivers to interact primarily through secure messaging (contact rates); and (2) willingness of caregivers to complete self-directed training (training completion rates).

Aim 2: Assess the feasibility and acceptability of the program from the payer perspective including: (1) average time spent per home-visit (including preparation and travel time); (2) average time per month spent responding to caregiver emails and coordinating care with primary care physicians; and (3 differences in face-to-face primary care, urgent care, and emergency department visit rates by PWD.

Aim 3: Test the hypotheses that (H1) caregiver participants in STAR-VTF will have lower levels of caregiver burden at 8 weeks and 6 months compared to an attention control group; and (H2) PWD participants in STAR-VTF will have lower rates of antipsychotic medication use at 6 months compared to control. Secondary outcomes are: caregiver depression and caregiver self-efficacy. The investigators propose to recruit 100 CG-PWD dyads (50 per arm).

This will be the first study to test a low intensity, self-directed caregiver training program with remote support from social workers. It will also be the first study to measure changes in antipsychotic medication use by PWD after caregiver training. Kaiser Permanente is an ideal setting because investigators have access to the complete electronic health record (EHR), prescription medication use, health care use, and demographic data. The investigators will be able to identify and enroll participants in real-time using an automated data "troll" as investigators have done previously. This study will be an important step in expanding access to training and support in a format that could be implemented within integrated delivery systems with capitated payments (i.e., Accountable Care Organizations). Growing use of EHR portals in these organizations will further increase demand for web-based care management/support. Demand will also increase as today's near-retirees, familiar with web-based applications, develop ADRD. Kaiser Permanente has pioneered such efforts and is the lead site in the Mental Health Research Network (MHRN). Findings from this study will inform a future multi-site pragmatic trial across the 13 health systems and 12 million enrollees in the MHRN.

ELIGIBILITY:
Current Criteria:

Investigators will identify and recruit Person with Dementia-Caregiver dyads in which the person with dementia has has made a healthcare visit in the last week where a diagnosis of Alzheimer's Disease or related dementia was recorded. Because we will enroll dyads, there are inclusion/exclusion criteria for both.

Participants

Persons with dementia inclusion criteria:

Aged ≥ 65 years Confirmed diagnosis of Alzheimer's Disease related disorders (ADRD) from the patient Electronic Health Record (EHR) or primary care physician KP members for a minimum of 180 days prior to the index visit date. Expected to live >= 6 months from enrollment

Persons with dementia exclusion criteria:

* A diagnosis of bipolar disorder or schizophreniform disorder
* The primary care physician's opinion is that the person with dementia is expected to live less than 6 months.
* Less that 65 years of age
* Primary language is not English (patient requires a translator).

Caregiver inclusion criteria:

* Aged ≥ 21 years
* Lives with person with dementia or within 8 miles
* Provides at least 8 hours of care per week
* Have access to a computer or other device where they can access MyChart, personal email, and websites to complete online training
* Use MyChart to email the doctors that care for the PWD they are caring for

Caregivers exclusion criteria:

* Diagnosis of Alzheimer's Disease or related disorders.
* Less than 21 years of age
* Are not the spouse, or adult child
* Unable to read and speak English
* Do not have access to a computer or other device where they can access MyChart, personal email, and websites to complete online training
* Do not use MyChart to email to doctors that care for the PWD they are caring for.

Previous Criteria:

Participants

The investigators will identify and recruit Person with Dementia-Caregiver dyads in which the person with dementia has filled a new prescription for an antipsychotic medication. Because we will enroll dyads, there are inclusion/exclusion criteria for both.

Persons with dementia inclusion criteria:

* Aged ≥ 65 years
* Diagnosis of Alzheimer's Disease related dementia (ADRD)
* A new prescription for an antipsychotic medication
* Living at home
* Expected to live >= 6 months from enrollment

Persons with dementia exclusion criteria:

* A diagnosis of bipolar disorder or schizophreniform disorder
* Living in an assisted living, skilled nursing facility, or memory facility
* The primary care physician's opinion is that the person with dementia is expected to live less than 6 months.

Caregiver inclusion criteria:

* Aged ≥ 21 years
* Lives with person with dementia or within 8 miles
* Provides at least 8 hours of care per week

Caregivers exclusion criteria:

* Diagnosis of Alzheimer's Disease or related disorders.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Dementia-Caregiver dyads were recruited based on whether the person with dementia had made a healthcare visit within the last week where a diagnosis of Alzheimer's Disease or related dementia was recorded between April 2020 and January 2023. The first dyad participants were enrolled in May 2020 and the last dyad was enrolled February 2023.
Pre-assignment Details: Using electronic health records, 935 patients with a dementia diagnosis were identified. After initial review of their electronic health record and contacting their provider for an opt out response, 592 fulfilled a subset of study inclusion criteria and their caregiver on file was contacted to assess further inclusion criteria. Of the 577 eligible dyad participants, 125 agreed to complete a phone screening for eligibility, with 67 dyads randomized and enrolled in the study.
Groups:
- Usual Care - Caregiver: Caregivers randomized to the usual care control condition will have one orientation phone visit with a coach and receive mailed material from the Alzheimer's Association, web links and template secure messages.
- Usual Care - Patient With Dementia: Patients with dementia randomized to the usual care control condition will be asked for consent to have their caregiver participate in the study and for the use of their medical record data.
- STAR-C VTF - Caregiver: Randomized Caregivers are offered:
  * A telephone orientation visit with a study coach to acquaint the caregiver to the 6-session STAR-VTF program and online learning environment.
  * A paper-based and electronic manual to identify priority behaviors, develop plans for addressing behaviors, and make plans for pleasant events.
  * 6 weekly telephone coaching visits lasting 30 minutes and corresponding to each of the 6 training modules.
  * Secure message (email) support within the patient portal, as needed, with the coach to help with personalizing the STAR-VTF curriculum for up to 6 months, as initiated by the caregiver.
- STAR-C VTF - Patient With Dementia: Patients with dementia randomized to the STAR-C VTF condition will be asked for consent to have their caregiver participate in the study and for the use of their medical record data.
Period: Overall Study
Arm/Group | Usual Care - Caregiver | Usual Care - Patient With Dementia | STAR-C VTF - Caregiver | STAR-C VTF - Patient With Dementia
Started (Surveys were only administered to caregiver participants in each arm.) | 32 | 32 | 35 | 35
Baseline Surveys (Surveys were only administered to caregiver participants in each arm.) | 31 | 0 (Patients with dementia did not complete any surveys. Surveys were only administered to the caregivers in both arms.) | 34 | 0 (Patients with dementia did not complete any surveys. Surveys were only administered to the caregivers in both arms.)
8-week Surveys (Surveys were only administered to caregiver participants in each arm.) | 20 | 0 (Patients with dementia did not complete any surveys. Surveys were only administered to the caregivers in both arms.) | 28 | 0 (Patients with dementia did not complete any surveys. Surveys were only administered to the caregivers in both arms.)
6-month Surveys (Surveys were only administered to caregiver participants in each arm.) | 18 | 0 (Patients with dementia did not complete any surveys. Surveys were only administered to the caregivers in both arms.) | 22 | 0 (Patients with dementia did not complete any surveys. Surveys were only administered to the caregivers in both arms.)
Completed | 18 | 0 (Patients with dementia did not complete any surveys. Surveys were only administered to the caregivers in both arms.) | 22 | 0 (Patients with dementia did not complete any surveys. Surveys were only administered to the caregivers in both arms.)
Not Completed | 14 | 32 | 13 | 35
Not completed — Death | 0 | 2 | 0 | 2
Not completed — Lost to Follow-up | 12 | 12 | 11 | 11
Not completed — Patient with Dementia Died | 2 | 0 | 2 | 0
Not completed — Patient with dementia were not administered surveys | 0 | 18 | 0 | 22

BASELINE CHARACTERISTICS:
Population: For this study, data collected from the the patients with dementia come from their electronic health record data. Caregivers were the focus of this study and the same measures were used for both arms. Measure descriptions clearly state which are from patients with dementia and caregivers, respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care - Caregiver | Usual Care - Patient With Dementia | STAR-C VTF - Caregiver | STAR-C VTF - Patient With Dementia | Total
Number analyzed (Participants) | 32 | 32 | 35 | 35 | 134
Age, Categorical [Count of Participants; unit: Participants] — Demographic data was collected from the patient with dementia's medical record and the caregiver demographic data was collected at a later date; we were not able to record all caregiver demographic data. Population: We collected the caregiver's demographic data at a later date for both arms; we have missing data for 10 caregivers in usual care and 8 caregivers in STAR-C VTF. The later collection date made it harder to reach participants that already completed the intervention, had withdrawn, or had completed the study. There is not a row to display missing data in this table.
  Participants
    number analyzed (Participants) | 22 | 32 | 27 | 35 | 116
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 3 | 0 | 8 | 0 | 11
    >=65 years | 19 | 32 | 19 | 35 | 105
Sex: Female, Male [Count of Participants; unit: Participants] — Demographic data was collected from the patient with dementia's medical record and the caregiver demographic data was collected at a later date; we were not able to record all caregiver demographic data. Population: We collected the caregiver's demographic data at a later date for both arms; we have missing data for 10 caregivers in usual care and 8 caregivers in STAR-C VTF. The later collection date made it harder to reach participants that already completed the intervention, had withdrawn, or had completed the study. There is not a row to display missing data in this table.
  Participants
    number analyzed (Participants) | 22 | 32 | 27 | 35 | 116
    Female | 18 | 14 | 17 | 17 | 66
    Male | 4 | 18 | 10 | 18 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Demographic data was collected from the patient with dementia's medical record and the caregiver demographic data was collected at a later date; we were not able to record all caregiver demographic data. Population: We collected the caregiver's demographic data at a later date for both arms; we have missing data for 10 caregivers in usual care and 8 caregivers in STAR-C. The later collection date made it harder to reach participants that already completed the intervention, had withdrawn, or had completed the study.
  Participants
    number analyzed (Participants) | 22 | 32 | 27 | 35 | 116
    Hispanic or Latino | 0 | 0 | 0 | 2 | 2
    Not Hispanic or Latino | 22 | 31 | 27 | 31 | 111
    Unknown or Not Reported | 0 | 1 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Demographic data was collected from the patient with dementia's medical record and the caregiver demographic data was collected at a later date; we were not able to record all caregiver demographic data. Population: We collected the caregiver's demographic data at a later date for both arms; we have missing data for 10 caregivers in usual care and 8 caregivers in STAR-C. The later collection date made it harder to reach participants that already completed the intervention, had withdrawn, or had completed the study.
  Participants
    number analyzed (Participants) | 22 | 32 | 27 | 35 | 116
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 1 | 1 | 0 | 2
    White | 22 | 29 | 26 | 33 | 110
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 2 | 0 | 2 | 4
Region of Enrollment [Number; unit: participants] — Demographic data was collected from the patient with dementia's medical record and the caregiver demographic data was collected at a later date. Although we were not able to collect all demographic data from the caregivers, all resided in the same region.
  participants
    United States | 32 | 32 | 35 | 35 | 67
Caregiver Mastery Scale [Mean (Standard Deviation); unit: units on a scale] — The Caregiver Mastery Scale is a 7-item self-report scale, indicating the extent to which respondents agree (5) or disagree (1) with each item. Three items with negative statements are reverse-scored. Total scores can range from 7 to 35, with higher scores reflecting greater caregiver mastery. This scale was only used with caregivers and were reported as the total score. Population: The Caregiver Mastery Scale is only completed by the caregiver.
  units on a scale
    number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    (all) | 20.5 (3.28) |  | 20.2 (3.37) |  | 20.3 (3.30)
Revised Memory and Problem Behavioral Checklist [Mean (Standard Deviation); unit: units on a scale] — Scale used to measure caregiver's observation of any memory or behavior issues over the past week. The potential range of the scale is 0-96 with higher scores reflecting more problems with memory or behaviors observed in the patient with dementia. This scale was only used with caregivers and were reported as the total score. Population: The Revised Memory and Problem Behavioral Checklist is only completed by the caregiver.
  units on a scale
    number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    (all) | 25.7 (16.38) |  | 30.5 (16.69) |  | 28.3 (16.54)
Kingston Caregiver Stress [Mean (Standard Deviation); unit: units on a scale] — This measure captures the caregiver's self-reported level of stress. Potential range of 10-50, with higher values indicating higher stress in the caregiver. This scale was only used with caregivers and were reported as the total score. Population: The Kingston Caregiver Stress is only completed by the caregiver.
  units on a scale
    number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    (all) | 23.6 (6.90) |  | 22.3 (6.57) |  | 22.9 (6.66)
RMBPC, Depression subscale [Mean (Standard Deviation); unit: units on a scale] — The Revised Memory and Behavior Problems Checklist, Depression subscale measure depression symptoms of the patient with dementia as reported by the caregiver. The sub scale range is 0-36; with a higher score indicating worse depression symptoms. Population: The RMBPC, Depression subscale is only completed by the caregiver.
  units on a scale
    number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    (all) | 7.3 (7.22) |  | 12.1 (11.94) |  | 10.1 (10.37)
Functional Activities Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Functional Activities Questionnaire measures the patient with dementia's dependency on their caregiver for daily activities as reported by the caregiver. Total range is 0-30; with a higher score indicating a higher dependence on the caregiver by the patient with dementia. Population: The Functional Activities Questionnaire is only completed by the caregiver.
  units on a scale
    number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    (all) | 22.0 (7.83) |  | 22.3 (5.23) |  | 22.2 (6.42)
Dementia Severity Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Dementia Severity Rating Scale measures the severity of dementia as observed by a caregiver in the patient with dementia. The subscale ranges are:
  A higher subscale score indicates worse dementia symptom.
  * Memory, Speech and Language, Ability to Get From Place to Place: range of 0-6
  * Recognition of Family Members, Social & Community Activity: range of 0-5
  * Orientation to Time, Place, Ability to Make Decisions, Home Activities & Responsibilities, Control of Urination and Bowels: range of 0-4
  * Personal Care - Cleanliness, Eating: range of 0-3 Population: The Dementia Severity Rating Scale is completed by the caregiver to report the patient with dementia's severity rating for each subscale.
  units on a scale
    Memory: number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    Memory | 3.96 (1.21) |  | 3.23 (1.38) |  | 3.54 (1.35)
    Speech & Language: number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    Speech & Language | 2.55 (1.47) |  | 2.27 (1.46) |  | 2.38 (1.46)
    Recognition of Family Members: number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    Recognition of Family Members | 1.40 (1.26) |  | 0.93 (0.98) |  | 1.13 (1.12)
    Orientation to Time: number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    Orientation to Time | 1.36 (0.79) |  | 1.30 (0.84) |  | 1.33 (0.81)
    Orientation to Place: number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    Orientation to Place | 1.55 (1.06) |  | 1.40 (1.10) |  | 1.46 (1.07)
    Ability to Make Decisions: number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    Ability to Make Decisions | 2.09 (0.92) |  | 2.50 (0.94) |  | 2.33 (0.94)
    Social & Community Activity: number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    Social & Community Activity | 2.59 (0.73) |  | 2.33 (0.92) |  | 2.44 (0.85)
    Home Activities and Responsibilities: number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    Home Activities and Responsibilities | 2.14 (1.08) |  | 2.37 (1.23) |  | 2.27 (1.10)
    Personal Care - Cleanliness: number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    Personal Care - Cleanliness | 1.14 (0.77) |  | 1.20 (0.81) |  | 1.17 (0.79)
    Eating: number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    Eating | 0.57 (0.75) |  | 0.43 (0.63) |  | 0.49 (0.67)
    Control of Urination and Bowels: number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    Control of Urination and Bowels | 1.36 (1.40) |  | 1.63 (1.35) |  | 1.52 (1.36)
    Ability to Get from Place to Place: number analyzed (Participants) | 32 | 0 | 35 | 0 | 67
    Ability to Get from Place to Place | 2.22 (1.30) |  | 2.20 (1.03) |  | 2.21 (1.14)

OUTCOME MEASURES:

1. Primary Outcome: Change in Caregiver Burden
Description: Self-reported caregiver burden assessed by the Disruption subscale on the Revised Memory and Behavior Problem Checklist (RMBPC) questionnaire. The range in subscale scores is 0 to 32 with higher scores representing a worse outcome.
Time Frame: Change from baseline caregiver burden at 6 months.
Population: We used multiple imputation on our entire sample of 67 caregivers, including baseline survey response, 8 week survey response, and 6 month survey response. As such, all individuals contributed information to the analyses.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Usual Care: Participants randomized to the control condition will have one orientation phone visit with a coach and receive mailed material from the Alzheimer's Association, web links and template secure messages.
- STAR-C VTF: Randomized Person Living With Dementia - Caregiver dyads are offered:
  * A telephone orientation visit with a study coach to acquaint the caregiver to the 6-session STAR-VTF program and online learning environment.
  * A paper-based and electronic manual to identify priority behaviors, develop plans for addressing behaviors, and make plans for pleasant events.
  * 6 weekly telephone coaching visits lasting 30 minutes and corresponding to each of the 6 training modules.
  * Secure message (email) support within the patient portal, as needed, with the coach to help with personalizing the STAR-VTF curriculum for up to 6 months, as initiated by the caregiver.
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 24.44 [19.69 to 29.20] | 22.30 [17.66 to 26.93]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.97, Regression, Linear

2. Secondary Outcome: Change in Caregiver Depression
Description: Self-reported caregiver depression assessed by the RMBPC, Depression subscale on the Revised Memory and Behavior Problem Checklist (RMBPC) questionnaire. The range in subscale scores is 0 to 36 with higher scores representing a worse outcome.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 7.80 [4.89 to 10.72] | 6.32 [3.88 to 8.76]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.55, Regression, Linear

3. Secondary Outcome: Change in Caregiver Self-efficacy
Description: Self-reported caregiver self-efficacy assessed by the Caregiver Mastery Scale. Total scores can range from 7 to 35, with higher scores reflecting greater caregiver mastery.
  The Caregiver Mastery Scale is a 7-item measure of self-efficacy. is a 7-item self-report scale, indicating the extent to which respondents agree (5) or disagree (1) with each item. Three items with negative statements are reverse-scored. Total scores can range from 7 to 35, with higher scores reflecting greater caregiver mastery.
Time Frame: Change from baseline caregiver mastery at 6 months.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 20.44 [19.22 to 21.64] | 21.42 [20.18 to 22.65]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.26, Regression, Linear

4. Secondary Outcome: Kingston Caregiver Stress Scale
Description: The Kingston Caregiver Stress Scale (KCSS) is designed to allow a family member (or other) caregiver to express his/her level of perceived stress, as it relates to caregiving. It can also be used to monitor changes in stress levels over time, as the caregiver's situation changes. Scores range from 10-50; a higher scores indicates higher levels of stress.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 22.13 [19.75 to 24.52] | 20.46 [18.19 to 22.72]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.42, Regression, Linear

5. Secondary Outcome: Number of Caregivers Who Responded to Surveys at 8-weeks
Description: We report the number of caregivers who completed their 8 week surveys by study arm.
Time Frame: 8 weeks from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
Participants | 20 | 28

6. Secondary Outcome: Number of Caregivers Who Responded to Surveys at 6-months
Description: We report the number of caregivers who completed their 6-month surveys by study arm.
Time Frame: 6 months from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
Participants | 18 | 22

7. Secondary Outcome: Number of Dyads Who Complete STAR-C VTF Online Training
Description: We will report completion rates by study arm at the end of the trial. Completion will be defined as completing 2 home-based visits, 1 phone-based visit and sending at least one secure message to a social worker in the baseline to 8-week period and one message in weeks 9 through 24.
Time Frame: 8 weeks from baseline
Population: We reviewed how many caregiver - patient with dementia dyads completed the 8 weeks of online STAR-C VTF separate from those that completed the week 8 follow-up surveys. We report on the number of dyads that completed the online training from the total number enrolled. The number differs from the participant flow form because some dyads did not complete the week 8 follow-up survey but did complete the online training.
Measure: Number; unit: dyads
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
dyads | 0 | 30

8. Secondary Outcome: Number of Inpatient Visits Had by Patient With Dementia
Description: Measured as the total number of inpatient visits had by patients with dementia within the study 6-month period.
Time Frame: End of follow-up (6 months)
Population: We analyzed our entire sample of 67 patients with dementia to understand how many touches they had with our care delivery system throughout the entire study. The total number differs from the participant flow as that is a reflection of completed follow-up surveys and not care delivery system touches.
Measure: Number; unit: Inpatient Visits
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
Inpatient Visits | 5 | 2

9. Secondary Outcome: Number of Primary Care Visits Had by Patient With Dementia
Description: Measured as the total number of primary care visits had by the patients with dementia within the study 6-month period.
Time Frame: End of follow-up (6 months)
Population: as for outcome 8
Measure: Number; unit: Primary Care Visits
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
Primary Care Visits | 22 | 30

10. Secondary Outcome: Number of Emergency Department Visits Had by Patient With Dementia
Description: Measured as the total number of emergency department visits had by patients with dementia within the study 6-month period.
Time Frame: End of follow-up (6 months)
Population: as for outcome 8
Measure: Number; unit: Emergency Department Visits
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
Emergency Department Visits | 13 | 17

11. Secondary Outcome: Antipsychotic Prescription Fills Rate for Patient With Dementia
Description: Average number of prescription fills for the patient with dementia after 8 weeks enrolled in the study. This data comes from the automated system pharmacy data.
Time Frame: After 8 weeks in the study
Population: We analyzed our entire sample of 67 patients with dementia to understand how many prescriptions were filled for the patient with dementia after 8 weeks in the study. The total number differs from the participant flow as that is a reflection of completed follow-up surveys and not prescription fills.
Measure: Mean (95% Confidence Interval); unit: Average number of prescription fills
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
Average number of prescription fills | 0.154 [0.030 to 0.228] | 0.031 [0.000 to 0.930]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.08, Regression, Linear

12. Secondary Outcome: Antipsychotic Prescription Refill Rate for Patient With Dementia
Description: Refill rates after initial medication dispensing, using automated system pharmacy data
Time Frame: 8 weeks after initial prescription
Population: We analyzed our entire sample of 67 patients with dementia to understand how many prescriptions were filled for the patient with dementia after 8 weeks in the study. The total number differs from the participant flow as that is a reflection of completed follow-up surveys and not prescription refills.
Measure: Mean (95% Confidence Interval); unit: Average number of prescription refills
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
Average number of prescription refills | .094 [0.000 to 0.200] | 0.114 [0.004 to 0.224]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.79, Regression, Linear

13. Secondary Outcome: Dementia Severity Rating Scale (DSRS) - Memory
Description: The Dementia Severity Rating Scale measures the severity of dementia as observed by a caregiver in the patient with dementia. The Memory subscale ranges from 0-6 and measures issues with memory. A higher subscale score indicates worse memory symptoms.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 4.05 [3.69 to 4.41] | 3.88 [3.51 to 4.26]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.60, Regression, Linear

14. Secondary Outcome: Dementia Severity Rating Scale (DSRS) - Speech and Language
Description: The Dementia Severity Rating Scale measures the severity of dementia as observed by a caregiver in the patient with dementia. The Speech and Language subscale ranges from 0-6 and measures issues with speech and language. A higher subscale score indicates worse ability to speak and converse with others.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 2.68 [2.13 to 3.25] | 2.68 [2.10 to 3.26]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.86, Regression, Linear

15. Secondary Outcome: Dementia Severity Rating Scale (DSRS) - Recognition of Family Members
Description: The Dementia Severity Rating Scale measures the severity of dementia as observed by a caregiver in the patient with dementia. The Recognition of Family Members subscale ranges from 0-5 and measures issues with recognition of family members. A higher subscale score indicates worse recognition of family members.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 1.10 [0.77 to 1.43] | 1.33 [0.99 to 1.67]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.46, Regression, Linear

16. Secondary Outcome: Dementia Severity Rating Scale (DSRS) - Orientation to Time
Description: The Dementia Severity Rating Scale measures the severity of dementia as observed by a caregiver in the patient with dementia. The Orientation to Time subscale ranges from 0-4 and measures issues with the patient with dementia's ability to orient themselves in time. A higher subscale score indicates worse ability to orient themselves in time.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 1.69 [1.33 to 2.05] | 1.62 [1.31 to 1.93]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.55, Regression, Linear

17. Secondary Outcome: Dementia Severity Rating Scale (DSRS) - Orientation to Place
Description: The Dementia Severity Rating Scale measures the severity of dementia as observed by a caregiver in the patient with dementia. The Orientation to Place subscale ranges from 0-4 and measures issues with the patient with dementia's ability to orient themselves. A higher subscale score indicates worse disorientation.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 1.92 [1.53 to 2.30] | 1.96 [1.61 to 2.31]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.63, Regression, Linear

18. Secondary Outcome: Dementia Severity Rating Scale (DSRS) - Ability to Make Decisions
Description: The Dementia Severity Rating Scale measures the severity of dementia as observed by a caregiver in the patient with dementia. The Ability to Make Decisions subscale ranges from 0-4 and measures issues with the patient with dementia's ability to make decisions for themselves. A higher subscale score indicates worse ability to make decisions for themselves.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 2.64 [2.32 to 2.97] | 2.47 [2.11 to 2.81]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.28, Regression, Linear

19. Secondary Outcome: Dementia Severity Rating Scale (DSRS) - Social & Community Activity
Description: The Dementia Severity Rating Scale measures the severity of dementia as observed by a caregiver in the patient with dementia. The Social & Community Activity subscale ranges from 0-5 and measures issues with the patient with dementia's ability to interact with those around them. A higher subscale score indicates worse ability to interact with others.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 2.62 [2.16 to 3.08] | 2.68 [2.40 to 2.97]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.82, Regression, Linear

20. Secondary Outcome: Dementia Severity Rating Scale (DSRS) - Home Activities & Responsibilities
Description: The Dementia Severity Rating Scale measures the severity of dementia as observed by a caregiver in the patient with dementia. The Home Activities & Responsibilities subscale ranges from 0-4 and measures issues with the patient with dementia's ability to do their usual things around the house. A higher subscale score indicates worse ability to complete home activities and responsibilities.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 2.91 [2.56 to 3.28] | 2.45 [2.17 to 2.72]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.04, Regression, Linear

21. Secondary Outcome: Dementia Severity Rating Scale (DSRS) - Personal Care - Cleanliness
Description: The Dementia Severity Rating Scale measures the severity of dementia as observed by a caregiver in the patient with dementia. The Personal Care - Cleanliness subscale ranges from 0-3 and measures issues with the patient with dementia's ability to take care of their personal hygiene independently. A higher subscale score indicates worse ability to maintain their cleanliness independently.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 1.36 [0.98 to 1.75] | 1.37 [1.09 to 1.64]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.98, Regression, Linear

22. Secondary Outcome: Dementia Severity Rating Scale (DSRS) - Eating
Description: The Dementia Severity Rating Scale measures the severity of dementia as observed by a caregiver in the patient with dementia. The Eating subscale ranges from 0-3 and measures issues with the patient with dementia's ability to eat independently. A higher subscale score indicates worse ability to eat independently.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 0.56 [0.28 to 0.84] | 0.83 [0.51 to 1.16]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.22, Regression, Linear

23. Secondary Outcome: Dementia Severity Rating Scale (DSRS) - Control of Urination and Bowels
Description: The Dementia Severity Rating Scale measures the severity of dementia as observed by a caregiver in the patient with dementia. The Control of Urination and Bowels subscale ranges from 0-4 and measures issues with the patient with dementia's ability to control their urination and bowels. A higher subscale score indicates worse ability to control their urination and bowels.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 1.94 [1.51 to 2.37] | 1.97 [1.58 to 2.37]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.85, Regression, Linear

24. Secondary Outcome: Dementia Severity Rating Scale (DSRS) - Ability to Get From Place to Place
Description: The Dementia Severity Rating Scale measures the severity of dementia as observed by a caregiver in the patient with dementia. The Ability to Get From Place to Place subscale ranges from 0-6 and measures issues with the patient with dementia's ability to get around on their own. A higher subscale score indicates worse ability to get around independently.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 2.43 [2.03 to 2.83] | 2.50 [2.16 to 2.84]
Statistical Analysis 1: Comparison: Usual Care vs STAR-C VTF; Test type: Other; p = 0.80, Regression, Linear

25. Other Pre Specified Outcome: Functional Activities Questionnaire (FAQ)
Description: The FAQ measures instrumental activities of daily living, such as preparing balanced meals and managing personal finances as observed by the caregiver in the patient with dementia. The tool consists of 10 questions with total scores ranging from 0-30. A minimum score of 9 indicates impaired functioning, and as the score increases from 9 indicating a greater reduction in functioning.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | STAR-C VTF
Number analyzed (Participants) | 32 | 35
units on a scale | 22.97 [20.76 to 25.17] | 24.34 [22.21 to 26.48]

ADVERSE EVENTS:
Time Frame: Each participant was assessed over the course of 6 months while they were in the study, from baseline to end of study.
Arm/Group | Usual Care - Caregiver | Usual Care - Patient With Dementia | STAR-C VTF - Caregiver | STAR-C VTF - Patient With Dementia
All-Cause Mortality (participants affected / at risk) | 0/32 | 2/32 | 0/35 | 2/35
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/35 | 4/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care - Caregiver (N=32) | Usual Care - Patient With Dementia (N=32) | STAR-C VTF - Caregiver (N=35) | STAR-C VTF - Patient With Dementia (N=35)
Hospitalization (General disorders) | 0 | NA | NA | 1
Mechanical Fall (Injury, poisoning and procedural complications) | 0 | NA | NA | 1
Difficulty Waking (Injury, poisoning and procedural complications) | 0 | NA | NA | 1
Distress (Psychiatric disorders) | 0 | NA | NA | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-08-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT04271046/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT04271046/SAP_001.pdf